CLINICAL TRIAL: NCT07207434
Title: Ability of VE818 to Reduce Enteropathogen Colonization and Improve Environmental Enteropathy in Pregnant Women: a Proof of Concept and Phase II Randomized Placebo-controlled Trial in Bangladesh, Pakistan, Zambia and Burkina Faso
Brief Title: Maternal Probiotic Intervention to Improve Gut Health-Trial II-Pakistan
Acronym: MPIGH-II
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); University of Zambia (Other); Institut Pasteur de Dakar (Other)
Responsible Party: Principal Investigator, Dr Syed Asad Ali, Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-9410-27780
Record Dates: First submitted 2025-08-16; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Environmental Enteric Dysfunction (EED); Stunting
Keywords: probiotic; microbiome; pregnant women; capscan device; urine LR; VE818; Pakistan; malnourished children; biomarkers; EED
MeSH Terms: conditions — Growth Disorders | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomisation will be carried out using sealed envelopes, using a randomisation code prepared by the trial statistician, which will be stratified by study centre. Each woman who gives Trial consent will be given a trial identification (TID) number, which will match the number on the randomisation envelopes.
  The trial will be blinded with an identical placebo. Samples will be run and analysed using TID only, with all data cleaning and re-assays carried out blinded. The trial statistician will unblind the lab data once the databases are finalised.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral vancomycin + VE818 (Active Comparator): Drug: VE818 VE818 is an 11-strain bacterial consortium rationally designed by Vedanta Biosciences Inc., to displace enteropathogens and reduce intestinal inflammation in pregnant women
  Drug: Oral Vancomycin Oral vancomycin in capsule form will be administered three times daily for 5 days at 250mg per dose. Because oral vancomycin is a non-absorbable antibiotic, the likelihood of systemic absorption is minimal and therefore, it is not associated with the adverse events attributable to the intravenous formulation
  Interventions: Drug: Oral Vancomycin; Drug: VE818
- Oral vancomycin + Placebo (Placebo Comparator): Drug: Placebo Enteric Capsules filled with approximately 400mg of Microcrystalline Cellulose (bulking agent)
  Drug: Oral Vancomycin Oral vancomycin in capsule form will be administered three times daily for 5 days at 250mg per dose. Because oral vancomycin is a non-absorbable antibiotic, the likelihood of systemic absorption is minimal and therefore, it is not associated with the adverse events attributable to the intravenous formulation
  Interventions: Drug: Oral Vancomycin; Drug: Placebo
- Observation only arm (No Intervention): The observational arm is a no-intervention control group within a Phase II randomized controlled trial that enrolls pregnant women colonized with at least 2 out of 11 selected bacterial enteropathogens recruited from community. This arm includes 48 participants per site (192 total across 4 sites) randomized in a 1:1:1 ratio alongside two intervention arms (oral vancomycin + placebo and oral vancomycin + VE818), with participants followed at comparable timepoints including baseline assessments, multiple visits during pregnancy, delivery, and up to 1 month postpartum for comprehensive evaluation of mother-infant dyads without receiving any study intervention.

INTERVENTIONS:
Drug: Oral Vancomycin — Oral vancomycin in capsule form will be administered three times daily for 5 days at 250mg per dose. Because oral vancomycin is a non-absorbable antibiotic, the likelihood of systemic absorption is minimal and therefore, it is not associated with the adverse events attributable to the intravenous formulation
  Arms: Oral vancomycin + Placebo; Oral vancomycin + VE818
Drug: VE818 — VE818 is an 11-strain bacterial consortium rationally designed by Vedanta Biosciences Inc., to displace enteropathogens and reduce intestinal inflammation in pregnant women.
  Arms: Oral vancomycin + VE818
Drug: Placebo — Enteric capsules filled with approximately 400mg of microcrystalline cellulose (bulking agent)
  Arms: Oral vancomycin + Placebo

SUMMARY:
Burden: Environmental Enteric Dysfunction (EED) is an enteropathic condition characterised by altered gut permeability, infiltration of immune cells, and changes in villous architecture and cell differentiation. EED is a major reason of malnourishment, poor neurological development, stunting, oral vaccine failure, and infection. It is believed that EED is responsible for 40% of all childhood stunting.

Relevance: This trial aims to investigate the concept that a probiotic or live biotherapeutic product, capable of improving gut microbiota composition, can also displace enteropathogens and reduce biomarkers of intestinal inflammation, thereby promoting gut health. This will restore healthy microbial signalling to the host epithelium, ameliorate barrier function through secretion of mucus and antimicrobial factors, and improve nutrient availability.

Objectives: The primary objective is to assess if administration of oral vancomycin followed by VE818 to pregnant women colonised with at least 2 out of 11 selected bacterial enteropathogens results in a significant change in the mean count of these organisms between the baseline and 2 weeks after completion of the intervention (Study Day 35d +2), compared to oral vancomycin followed by placebo.

Methods: Pregnant women will be recruited from the community of Matiari in Pakistan. The study population will be women aged 18 years or older in the first trimester or early second trimester of pregnancy. Study procedures will be explained in detail, and written consent will be taken before enrollment. Those women who give consent to participation will undergo a screening process, which will check if any exclusion criteria are fulfilled. After consent and screening, they will be randomised into one of the three arms: intervention arm (oral vancomycin followed by VE818), placebo-control arm (oral vancomycin followed by placebo), or observation-only arm. The allocation sequence will be generated by the trial statistician using a code with block permutation. The participant will remain free to withdraw at any time from the trial without giving reasons and without prejudicing her further treatment. Biological samples, including blood, saliva, urine, stool, vaginal swab, and intestinal luminal contents through CapScan. CapScan is a non-invasive device (capsule) that collects gastrointestinal samples along the gastrointestinal tract following ingestion and passes into the stool.

Outcome measures/variables: The primary endpoint is the change in the mean count in the number of 11 selected fecal bacterial pathogen groups present between baseline and 2 weeks after completion of the 14-day course with Placebo or VE818 (Study arms 2 and 3), which corresponds to the 35th day, +2 from the first dose of oral vancomycin.

The 11 enteropathogen targets will be detected by customized real-time quantitative PCR-based TaqMan Array Cards (TAC-qPCR) and include the following organisms: Aeromonas, Campylobacter coli, Campylobacter jejuni, Campylobacter Pan, Enteroaggregative Escherichia coli (E. coli), Enteropathogenic E. coli, Enterotoxigenic E. coli, Plesiomonas, Shigella_Enteroinvasive E. coli (EIEC), Salmonella, and Klebsiella pneumoniae

DETAILED DESCRIPTION:
A total of 144 pregnant women in their second trimester will be enrolled. Subsequently, 96 will be randomized to receive an antibiotic for 5 days, followed by a 1-day washout period (1 week), and then either a probiotic or a placebo for 2 weeks. It will be a double-blind trial.

Pregnant women will be recruited in the community through a demographic surveillance system established in Matiari, Pakistan. The study staff will approach the potential participants and will introduce them to this study. If Participants agree, a screening consent form will be administered. During this, investigators will conduct a clinical assessment and measure the participants' hemoglobin levels. Additionally, a gestational ultrasound will be performed to confirm the trimester/gestational weeks, and a stool TAC will be collected to detect the presence of enteropathogens. Based on the screening results and clinical staff assessment, women will be enrolled after giving their consent to participate in the trial.

Once the participant is enrolled, investigators will collect blood, urine, LR, Vaginal Swab, and stool samples (flash frozen and CapScan) before giving them antibiotics and then either a placebo or probiotic (which will be replenished daily).

Investigators will then follow them daily for compliance and adverse event data collection for both antibiotic and then either a placebo or probiotic for 21 days (3 weeks). Investigators will collect blood, urine, LR, Vaginal Swab, and stool samples (flash frozen and CapScan) after completing the intervention.

The investigator will also conduct interval visits at different timepoints. Gestational ultrasounds, BIA, Skinfold, and Anthropometry will be performed at screening at 16, 20, 24, 28, 32, and 36 weeks of gestation.

Pregnancy outcomes will be recorded, and then the 1-month post-birth follow-up of mother and child will be done for anthropometry and morbidity data collection.

ELIGIBILITY:
Inclusion criteria

* Women aged 18 years or older in their first or early second trimester of pregnancy (13-17 weeks of gestational age [GA]), living in defined geographical areas of Bangladesh (Matlab), Pakistan, Zambia, and Burkina Faso, where it can be assumed that environmental enteropathy is prevalent
* Presence of any 2 out of 11 selected bacterial pathogen targets (Aeromonas, Campylobacter coli, Campylobacter jejuni, Campylobacter Pan, Enteroaggregative Escherichia coli, Enteropathogenic Escherichia coli, Enterotoxigenic Escherichia coli, Plesiomonas, Shigella_EIEC, Salmonella and Klebsiella pneumoniae in fecal samples measured by TAC-qPCR.
* Presence of any of the following WASH conditions -

  1. use surface water, unimproved water, or limited water for drinking; OR
  2. use surface water, unimproved water, or limited water for cooking; OR
  3. use surface water, unimproved water, or limited water for washing utensils; OR
  4. practice open defecation, use unimproved sanitation (toilet facility), or limited sanitation (toilet facility); OR
  5. lack facility or have limited facility for handwashing

Exclusion criteria

Potential participants will not be enrolled if they:

* have MUAC ≥30 cm
* are carrying more than one fetus (i.e., multiple pregnancy)
* have diarrhea, defined as the passage of three or more loose stools per 24 hours, or have had diarrhea in the preceding 14 days
* have fever or an active infection
* have taken antibiotics or probiotics in the preceding 14 days
* have taken steroids or non-steroidal anti-inflammatory drugs in the preceding 14 days
* have severe anemia as determined using finger stick Hb < 8 g/dl
* have a history of chronic digestive disease
* have any gastrointestinal contraindication to ingestion of a capsule (known or suspected gastrointestinal obstruction, stricture, fistula, gastroparesis, or any swallowing disorder)
* have known immunocompromised status (known history of HIV infection, autoimmune disease, diabetes mellitus, etc.)
* have known drug hypersensitivity/allergy/intolerance
* have chronic disease or any other illness or condition which in the opinion of the investigator will complicate the assessment of safety or efficacy
* are medically disqualified: Any potential participant who is deemed medically unfit for trial enrollment by a non-study healthcare provider, due to the presence of severe or unstable health conditions that could compromise safety or interfere with the study outcomes, will be excluded from participation
* have a plan to observe fast any time during the intervention period
* have a plan to leave the study area within the follow-up period
* are participating in any other interventional trial
* belong to a household from which another woman is already enrolled in the study
* but may be enrolled if/when these disqualifiers have expired.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All pregnant women in their first or early second trimester of pregnancy, residing in the Matiari district, who meet the eligibility criteria described below.
Enrollment: 144 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Mean Count of 11 Selected Fecal Bacterial Pathogen Groups as Measured by TAC-qPCR between enrollment and 2 weeks after completion of the 14-day course with Placebo or VE818 | Between enrollment and 2 weeks after completion of the 14-day course with Placebo or VE818
  The primary endpoint is the change in the mean count in the number of 11 selected fecal bacterial pathogen groups present between enrollment and 2 weeks after completion of the 14-day course with Placebo or VE818 (Study arms 2 and 3), which corresponds to 35th day, +2 from the first dose of oral vancomycin.

SECONDARY OUTCOMES:
Change in prevalence of specific enteropathogens not included in the primary endpoint in pregnant women as Measured by TAC-qPCR | Enrollment, Day 6 (18 weeks gestation), Day 21, Day 35 (23 weeks gestation), Day 63 (28 weeks gestation), and 7 days post-partum.
  Change in prevalence of specific enteropathogens (i.e., rotavirus, norovirus, Giardia, Cryptosporidium, and bacterial pathogens not included in the primary endpoint) in pregnant women detected in feces by TAC-qPCR between baseline (Day 0), end of oral vancomycin treatment (Day 6) the last dose of the 14-day VE818 intervention (21st day, +2), 14 days after the last dose of VE818 (35th day, +2), 42 days after the last dose of VE818 (63rd day, +2), and 7 day post-partum in the Treatment arm compared to Placebo arm and Observation-only arm.
Engraftment of VE818 strains in pregnant women as Measured by Shotgun Metagenomic Sequencing | At Day 21, Day 35 (23 weeks gestation), Day 63 (28 weeks gestation), and 7 days post-partum.
  Engraftment of VE818 strains in pregnant women as measured by shotgun metagenomic sequencing of fecal samples collected at the end of the 14-day VE818 intervention (21st day, +2), 14 days after the last dose of VE818 (35th day, +2), 42 days after the last dose of VE818 (63rd day, +2) and 7 days post-partum
Change from Enrollment in the Concentration of a Panel of Plasma Biomarkers as Measured by ELISA | At Enrollment, Day 6 (18 weeks gestation), Day 35 (23 weeks gestation), and Day 63 (28 weeks gestation).
  Change in a panel of plasma biomarkers (CRP, AGP, sCD14, LBP, CD163 and iFABP) in pregnant women as measured by ELISA between baseline (Day 0), end of oral vancomycin treatment (Day 6), 14 days after the last dose the of 14-day intervention (35th day, +2) and, 42 days after the last dose of VE818 (63rd day, +2) in the Treatment arm compared to Placebo arm and Observation-only arm.
Change from Enrollment in the Concentration of a Panel of Fecal Biomarkers as Measured by ELISA | At Enrollment, Day 6 (18 weeks gestation), Day 21, Day 35 (23 weeks gestation), Day 63 (28 weeks gestation), and 7 days post-partum
  Change in a panel of fecal biomarkers (myeloperoxidase, neopterin, calprotectin and lipocalin) in pregnant women as measured by ELISA between baseline (Day 0) , end of oral vancomycin treatment (Day 6), the last dose of the 14-day VE818 intervention (21st day, +2), 14 days after the last dose of VE818 (35th day, +2) 42 days after the last dose VE818 (63rd day, +2), and 7 day post-partum in the Treatment arm, compared to Placebo arm and Observation-only arm.
Change from Enrollment in Intestinal Permeability as Measured by Lactulose/Rhamnose (LR) Ratio | At Enrollment and Day 35 (23 weeks gestation).
  Change in intestinal permeability as measured by Lactulose/Rhamnose (LR) ratio in pregnant women between baseline and 14 days after the last dose of 14-day VE818 intervention (35th day, +2) in the Treatment arm, compared to Placebo arm and Observation-only arm.
Change from Enrollment in Alpha and Beta Diversity of Fecal Microbiome as Measured by Shotgun Metagenomics Sequencing | At Enrollment, Day 6 (18 weeks gestation), Day 21, Day 35 (23 weeks gestation), Day 63 (28 weeks gestation), and 7 days post-partum.
  Change in alpha and beta diversity of fecal microbiome in pregnant women as measured by shotgun metagenomics sequencing between baseline (Day 0), end of oral vancomycin treatment (Day 6), the last dose of the 14-day VE818 intervention (21st day, +2), 14 days after the last dose of VE818 (35th day, +2 day), 42 days after the last dose of VE818 (63rd day, +2), and 7 day post-partum in the Treatment arm, compared to Placebo arm and Observation-only arm
Change from Enrollment in Alpha and Beta Diversity of Vaginal Microbiome as Measured by Shotgun Metagenomics Sequencing | At Enrollment, Day 6 (18 weeks gestation), Day 35 (23 weeks gestation), and Day 63 (28 weeks gestation).
  Change in alpha and beta diversity of vaginal microbiome in pregnant women as measured by shotgun metagenomics sequencing between baseline, end of oral vancomycin treatment (Day 6), 14 days after the last dose of the 14-day VE818 intervention (35th day, +2), and 42 days after the last dose of VE818 (63rd day, +2), in the Treatment arm, compared to Placebo arm and Observation-only arm
Change from Enrollment in Alpha and Beta Diversity of Oral Microbiome as Measured by Shotgun Metagenomics Sequencing | At Enrollment and Day 35 (23 weeks gestation).
  Change in alpha and beta diversity of oral microbiome in pregnant women as measured by shotgun metagenomics sequencing between baseline (Day 0) (and 14 days after the last dose of the 14-day VE818 intervention (35th day, +2), in the Treatment arm, compared to Placebo arm and Observation-only arm
Change from Enrollment in the Metabolomic Profile of Plasma and Stool Samples | At Enrollment, Day 6 (18 weeks gestation), Day 21 (stool only), Day 35 (23 weeks gestation), Day 63 (28 weeks gestation), and 7 days post-partum (stool only).
  Change in metabolome (plasma, and stool) in pregnant women between baseline (Day 0), end of oral vancomycin treatment (Day 6), the last dose of the 14-day VE818 intervention (21st day +2; stool only), 14 days after the last dose of VE818 (35th day+2) 42 days after the last dose of VE818 (63rd day +2) and 7 days post birth (stool only) in the Treatment arm, compared to Placebo arm and Observation-only arm

OTHER OUTCOMES:
Difference in the rate of weight gain during the second and third trimester of pregnancy | Second (13 to 28 weeks of gestation) and third trimester of pregnancy (28 to 40 weeks of gestation)
  Difference in the rate of weight gain during the second and third trimester of pregnancy between Treatment arm and Placebo and Observation-only arms
Difference in fetal growth trajectories | At gestational weeks 16, 20, 24, 28, 32, and 36
  Difference in fetal growth trajectories as measured by serial ultrasound evaluation of intrauterine growth between Treatment arm and Placebo and Observation-only arms
Difference in placental insufficiency | At gestational weeks 28, 32, and 36
  Difference in placental insufficiency as measured by ultrasound-derived cerebroplacental ratio (CPR) between Treatment arm and Placebo and Observation-only arms
Difference in placental stress | First (up to 13 weeks of gestation), second (14 to 28 weeks of gestation), and third trimester of pregnancy (28 to 40 weeks of gestation)"
  Difference in placental stress measured through sFlt-1/PlGF ratio between Treatment arm and Placebo and Observation-only arms
Change from Enrollment in Alpha and Beta Diversity in the Gut Microbiota of Pregnant Women as Measured by Shotgun Metagenomic Sequencing of CapScan Samples | Enrollment and Day 35 (23 weeks gestation)
  Change in alpha and beta diversity in the gut microbiota of pregnant women as measured by shotgun metagenomic sequencing of intestinal fluid obtained using CapScan between baseline and 14 days after the last dose of the 14-day VE818 intervention (35th day, +2), in the Treatment arm, compared to Placebo arm and Observation-only arm
Engraftment of VE818 Strains in CapScan Samples as Measured by Shotgun Metagenomic Sequencing | Enrollment and Day 35 (23 weeks gestation)
  Engraftment of VE818 strains in CapScan samples collected 14 days after the last dose of VE818 (35th day, +2) as measured by shotgun metagenomic sequencing
Difference in Average Count of Enteropathogens in Infants as Measured by TAC-qPCR | 7 days post birth
  Difference in average count of enteropathogens in infants detected in feces by TAC-qPCR 7 days after birth between Treatment arm and Placebo and Observation-only arms
Difference in Concentration of a Panel of Fecal Biomarkers in Infants as Measured by ELISA | 7 days post birth
  Difference in a panel of fecal biomarkers (myeloperoxidase, neopterin, calprotectin and lipocalin) in infants as measured by ELISA 7 days after birth between Treatment arm and Placebo and Observation-only arms
Difference in Alpha and Beta Diversity of Fecal Microbiome in Infants as Measured by Shotgun Metagenomics Sequencing | 7 days post birth
  Difference in alpha and beta diversity of fecal microbiome in infants as measured by shotgun metagenomics sequencing 7 days after birth between Treatment arm and Placebo and Observation-only arms
Detection of VE818 Organisms in Infants as Measured by Metagenomic Analysis | 7 days post birth
  Detection of VE818 organisms in infants measured via metagenomic analysis of fecal samples collected 7 days after birth
Difference in Fecal Metabolomic Profile in Infants | 7 days post birth
  Difference in fecal metabolome in infants 7 days after birth between Treatment arm, Placebo arm and Observation-only arms
Variability in Endpoint Assays Across Geographies and Laboratories as Measured by Coefficient of Variation Analysis | At Enrollment, Day 6 (18 weeks gestation), Day 21, Day 35 (23 weeks gestation), Day 63 (28 weeks gestation), and 7 days post-partum.
  Variability in endpoint assays across geographies and laboratories
Difference in Perinatal Outcomes as Measured by Standardized Clinical Assessment | From 20 weeks gestation through 7 days post-birth
  Difference in perinatal outcomes between Treatment arm, Placebo arm and Observation-only arms
Difference in Birth Anthropometry as Measured by Standard Clinical Measurements (Weight, Length, Head Circumference) | At birth
  Difference in birth anthropometry between Treatment arm, Placebo arm and Observation-only arms
Difference in Infant Growth Measures as Assessed by Standard Anthropometric Measurements | 1 month post birth
  Differences in growth measures of the infants 1 month post birth between Treatment arm, Placebo arm and Observation-only arms
Difference in women's postpartum weight change | 1 month post-partum
  Differences in women's postpartum weight change (loss/retention) between Treatment arm, Placebo arm and Observation-only arms
Difference in Maternal Immune Responses as Measured by Cytokine Analysis and Immunological Assays | At Enrollment, Day 6 (18 weeks gestation), Day 21, Day 35 (23 weeks gestation), Day 63 (28 weeks gestation), 7 days post-partum. and 1 month post-partum
  Differences in maternal immune responses in plasma, cord blood and breast milk between Treatment arm, Placebo arm and Observation-only arms
Difference in Gene Expression in Maternal and Infant Stool Samples as Measured by RNA Sequencing Analysis | At Enrollment, Day 6 (18 weeks gestation), Day 21, Day 35 (23 weeks gestation), Day 63 (28 weeks gestation), and 7 days post-partum.
  Differences in gene expression in maternal and infant stool samples between Treatment arm, Placebo arm and Observation-only arms
Difference in Infant Morbidity as Assessed by Clinical Evaluation and Medical Record Review | 1 month post birth
  Infant Morbidity as Assessed by Clinical Evaluation and Medical Record Review

CONTACTS AND LOCATIONS:
Overall Officials: Asad Ali Syed, MPH, Principal Investigator — Aga Khan University
Locations (1):
- Mother and Child Health Research and Training Center, AKU, Matiari, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 24 months of study completion.
Access Criteria: Data access requests will be reviewed by the Trial Management Group. Requestors will be required to sign a Data Access Agreement.